CLINICAL TRIAL: NCT00723294
Title: A Phase II Trial Exploring the Success of Cryoablation Therapy in the Treatment of Invasive Breast Carcinoma
Brief Title: Cryoablation Therapy in Treating Patients With Invasive Ductal Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z1072; CDR0000600976
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; male breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Breast Neoplasms, Male | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cryoablation) (Experimental): A cryoprobe is inserted percutaneously under ultrasound guidance into the targeted lesion. Patients undergo ablation using a freeze-thaw-freeze cycle lasting approximately 6-10-6 or 8-10-8 minutes, respectively. Patients undergo surgical resection and sentinel lymph node biopsy and/or axillary dissection within 28 days after completion of cryoablation. Patients complete the Brief Pain Inventory before and after cryoablation and after surgery.
  Interventions: Procedure: cryosurgery; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: cryosurgery
Procedure: therapeutic conventional surgery

SUMMARY:
This phase II trial is studying how well cryoablation therapy works in treating patients with invasive ductal breast cancer. Cryoablation kills tumor cells by freezing them. This may be an effective treatment for patients with invasive ductal breast cancer.

DETAILED DESCRIPTION:
This is a phase II non-randomized exploratory study. All fully eligible and registered patients will undergo imaging by mammography, ultrasound, and breast MRI. Patients will then undergo complete surgical resection of the primary tumor. The primary and secondary objectives of the study are described below.

OBJECTIVES:

Primary

* To determine the rate of complete tumor ablation in patients treated with cryoablation, with complete tumor ablation defined as no remaining invasive or in situ carcinoma present upon pathological examination of the targeted lesion

Secondary

* To evaluate the negative predictive value of MRI in the post-ablation setting to determine residual in situ or invasive breast carcinoma
* To describe the adverse events associated with cryoablation
* To prospectively gather pain assessment data on cryoablation and surgical resection
* Explore technical variables that may affect the success of cryoablation

ELIGIBILITY:
1. Unifocal primary invasive ductal breast carcinoma diagnosed by core needle biopsy. NOTE: Patients with lobular carcinoma, multifocal and/or multicentric ipsilateral breast cancer, multifocal calcifications, or DCIS with microinvasion are NOT eligible. Patients with contralateral disease will remain eligible.
2. No history of en bloc open surgical biopsy and/or lumpectomy for diagnostic/treatment of the index breast cancer. Note: Prior rotational and/or vacuum-assisted core biopsies are permitted if no significant distortion is seen on imaging that could obscure visualization and detection of residual disease on MRI, or visualization of cancer on ultrasound for cryoablation procedure.
3. Tumor size ≤ 2.0 cm in greatest diameter. Specifically, the tumor must measure ≤ 2.0 cm in the axis parallel to the treatment probe and ≤ 1.5 cm in the axis anti-parallel to the treatment probe. Largest size measured by required scans (mammogram, ultrasound and MRI) will be used to determine eligibility.
4. Tumor enhancement on pre-study MRI.
5. Tumor with < 25% intraductal components in the aggregate. NOTE: The percent intraductal component from the patient's diagnostic biopsy must be available prior to registration. If the biopsy pathology report does not contain the percent intraductal component, then re-review of pathology slides and creation of a report addendum or note-to-file by the reviewing pathologist will be required.
6. No prior or planned neoadjuvant chemotherapy for breast cancer.
7. Non-pregnant and non-lactating. Patients of childbearing potential must have a negative serum or urine pregnancy test. NOTE: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential.
8. Adequate breast size for safe cryoablation. Male breast cancer patients and female breast cancer patients with breasts too small to allow safe cryoablation are not eligible as the minimal thickness of the breast tissue does not lend itself to cryoablation. NOTE: For patients with breast implants, the treating physician must document that adequate distance exists between the lesion and the implant to ensure that the ablated lesion will not contact or jeopardize the implant.
9. Patients with prior in-situ or invasive breast carcinomas are eligible if the prior carcinomas occurred in the contralateral breast. Patients with prior in-situ or invasive carcinomas of the ipsilateral breast are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rache M. Simmons, MD, Study Chair — Weill Medical College of Cornell University
Locations (16):
- United States (16):
  - Providence Saint Joseph Medical Center, Burbank, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - University of South Florida College of Medicine, Tampa, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Hospital/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Bethesda North Hospital, Cincinnati, Ohio
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Bellingham Breast Center, Bellingham, Washington

REFERENCES:
- [Result] Simmons RM, Ballman KV, Cox C, Carp N, Sabol J, Hwang RF, Attai D, Sabel M, Nathanson D, Kenler A, Gold L, Kaufman C, Han L, Bleznak A, Stanley Smith J, Holmes D, Fornage B, Le-Petross C, Hoda S, McCall L, Hunt KK; ACOSOG investigators. A Phase II Trial Exploring the Success of Cryoablation Therapy in the Treatment of Invasive Breast Carcinoma: Results from ACOSOG (Alliance) Z1072. Ann Surg Oncol. 2016 Aug;23(8):2438-45. doi: 10.1245/s10434-016-5275-3. Epub 2016 May 24. PMID 27221361

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cryoablation): A cryoprobe is inserted percutaneously under ultrasound guidance into the targeted lesion. Patients undergo ablation using a freeze-thaw-freeze cycle lasting approximately 6-10-6 or 8-10-8 minutes, respectively. Patients undergo surgical resection and sentinel lymph node biopsy and/or axillary dissection within 28 days after completion of cryoablation.
Period: Overall Study
Arm/Group | Treatment (Cryoablation)
Started | 99
Completed | 86
Not Completed | 13
Not completed — Lobular histology | 2
Not completed — >25% intraductal component | 1
Not completed — No MRI tumor enhancement | 1
Not completed — 1.0-Tesla MRI | 1
Not completed — No cryoabalation | 2
Not completed — Did not undergo surgery | 1
Not completed — Treated prior to registration | 1
Not completed — Treated by non-credentialed surgeon | 1
Not completed — Benign lesion | 1
Not completed — Withdrawal by Subject | 1
Not completed — No treatment due to probe failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cryoablation)
Number analyzed (Participants) | 86
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Tumor Ablation
Description: The primary endpoint for this study is the rate of complete ablation. Complete ablation is defined as no remaining invasive or in situ carcinoma present upon pathological examination of the targeted lesion. The rate (percentage) will be computed as the number of patient lesions with complete tumor ablation divided by the total number of eligible patient lesions. This rate will be estimated by the binomial point estimate (number of patients with no pathological evidence of residual disease in the targeted lesion after ablation divided by the number of eligible patients) and a one-sided 90% binomial confidence interval (interval with a lower bound).
Time Frame: Up to 14 days post surgery
Population: One patient had bilateral disease and therefore outcomes are reported for 87 lesions.
Measure: Number (90% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Treatment (Cryoablation)
Number analyzed (Participants) | 86
Number analyzed (lesions) | 87
percentage of lesions | 75.9 [67.1 to 83.2]

2. Secondary Outcome: Negative Predictive Value of MRI
Description: Negative predictive value of MRI: The negative predictive rate of MRI will be estimated as the number of patients with no residual disease upon pathologic review of the resected tissue AND with a MRI that indicated no residual disease divided by the number of patients who had an MRI that indicated no residual disease. Both a binomial point estimate and 90% two-sided confidence interval will be computed.
Time Frame: Up to 14 days post cryoablation
Population: One patient had bilateral disease and therefore outcomes are reported for 87 cancers.
Measure: Number (90% Confidence Interval); unit: percentage of cancers
Units Other Than Participants: cancers
Arm/Group | Treatment (Cryoablation)
Number analyzed (Participants) | 86
Number analyzed (cancers) | 87
percentage of cancers | 81.2 [71.4 to 88.8]

3. Secondary Outcome: Adverse Events
Time Frame: Up to 14 days post surgery
Reporting Status: Not Posted, anticipated posting 2017-12

4. Secondary Outcome: Pain Assessment
Time Frame: Up to 14 days post surgery
Reporting Status: Not Posted, anticipated posting 2017-12

ADVERSE EVENTS:
Time Frame: Adverse events are assessed 14 to 28 days post-cryoablation and within 14 days post surgery.
Description: Toxicities/adverse events must be described and graded using the terminology and grading categories defined in the most current version of the NCI's Common Toxicity Criteria (CTCAE) version 3.0. NOTE: CTCAE Version 3 will continue to be used for determining dose modifications/delays and for routine adverse event reporting. Effective October 1, 2010, CTCAE Version 4 will be used for expedited adverse event reporting only.
Arm/Group | Treatment (Cryoablation)
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 48/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cryoablation) (N=90)
Lymphatic disorder (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 6 (7)
Pain (General disorders) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 33 (47)
Intraoperative breast injury (Injury, poisoning and procedural complications) | 1 (2)
Seroma (Injury, poisoning and procedural complications) | 8 (8)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 32 (45)
Nipple deformity (Reproductive system and breast disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes